CLINICAL TRIAL: NCT02008058
Title: LCCC 1231: Observational Longitudinal Study of Pain in Men With Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Observational Longitudinal Study of Pain in Men With Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Memorial Sloan Kettering Cancer Center (Other); Johns Hopkins University (Other); University of Washington (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1231; 12-2562 (Other: UNC IRB)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Castrate-Resistant Prostate Cancer
Keywords: Metastatic Castrate-Resistant Prostate Cancer; LCCC 1231; Lineberger Comprehensive Cancer Center; UNC Lineberger; Prostate Cancer; Pain
MeSH Terms: conditions — Prostatic Neoplasms; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single Arm: Surveys, diaries, clinical assessments of men with metastatic castrate-resistant prostate cancer
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Patients will report pain and analgesic use through the automated telephone system, for 7 days in a row, once every 6 weeks. Data from diagnostic tests (CT Abdomen/Pelvis, Bone Scan, PSA, and circulating tumor cells) conducted during the study period will be collected from medical records by local personnel and entered into the secure online database quarterly, but no specific tests or schedules will be required in this observational study. Patients will remain on study for up to 26 months (slightly longer than the expected median survival in this population based on data from docetaxel, abiraterone, and MDV3100 pivotal phase 3 trials).
  Other Names: Webcore telephone survey system

SUMMARY:
This is a single-arm observational longitudinal study in of patients with metastatic castrate-resistant prostate cancer designed to assess the longitudinal trajectory of pain and other symptoms.

DETAILED DESCRIPTION:
This is a single-arm observational longitudinal study in of patients with metastatic castrate-resistant prostate cancer designed to assess the longitudinal trajectory of pain and other symptoms. The study aims to address several key methodological questions that will inform the design of future clinical trials with symptom endpoints in this population, including: the definition of "clinically meaningful" pain; criteria for concluding a clinically meaningful pain reduction; criteria for concluding clinically meaningful pain progression; reliable methods quantifying analgesic use (given that "equianalgesic tables" and "point scoring systems" are generally considered unreliable by pain researchers and regulatory agencies , , ); ideal recall periods for pain questions; tradeoffs of different frequencies of symptom reporting; symptom trajectories over time; and associations of pain scores with other metrics used in prostate cancer research (imaging, PSA values, circulating tumor cells, etc).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be ≥ 18 years old on the day of consent.
* The subject is able to understand written and spoken English
* The patient must have histologically or cytologically confirmed prostate adenocarcinoma.
* The subject must have castration-resistant prostate cancer (CRPC)
* The subject must have metastatic disease involving bone, seen on radiographic imaging (bone scan, CT scan, PET scan, or MRI).
* The subject must be in a castrate state (e.g., currently receiving androgen deprivation therapy or have had an orchiectomy).
* The subject must be starting any line treatment post-androgen deprivation/antiandrogen therapy, such as the following: chemotherapy (e.g., docetaxel, paclitaxel, carboplatin, cabazitaxel, or mitoxantrone); abiraterone acetate; MDV3100; ketoconazole; sipuleucel-T; Radium 223.
* The subject owns or has regular access to a telephone (cellular or land line).
* The subject is willing and able to self-report pain and analgesic use via an automated telephone system.
* The subject is willing and able to provide informed consent.

Exclusion Criteria:

* The subject has small cell or predominantly neuroendocrine differentiated prostate tumor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of pain palliation responders | 6 weeks
  Determine the proportion of pain palliation responders and the proportion experiencing pain progression will be presented along with 95% confidence intervals.

SECONDARY OUTCOMES:
Clinical significance of pain score changes | 6 weeks
  Determine the clinical significance of pain score changes. Pain score changes will be compared with each of the following "anchors": patient rating of change in pain, as well as changes in patient functional status, analgesic use, and various measures of disease status (imaging, PSA, circulating tumor cells). ROC curves derived using logistic regression analyses will be used to characterize the association between change in pain scores and clinically important improvement (defined by anchor variables).
Prevalence and trajectory of pain progression and pain palliation | 3 weeks
  Descriptive statistics, including Kaplan-Meier, will be used to report findings for the proportion of asymptomatic men who ultimately develop pain, the median time until asymptomatic men develop pain, the median time until men with pain experience pain progression, and the median time until men with pain experience pain palliation.
Quantifying analgesic medication use | 26 months
  Three different approaches to calculating a single value to represent total analgesic use will be compared: 1) equianalgesic tables published in guidelines of the National Comprehensive Cancer Network (NCCN) which convert various drugs and doses to "morphine equivalents"; 2) point scoring systems used in prior pivotal phase 3 trials based on the World Health Organization analgesic ladder in which lower points are assigned to weaker agents/doses and vice versa for stronger agents/doses; and 3) individual drug dose quantification, a dose recently suggested by the FDA but never empirically evaluated, in which each analgesic is considered individually and a 25% change in dose is considered an increase or decrease for each.
Frequency of pain reporting | 7 days
  Seven consecutive days of reporting a pain item with a 24-hour recall item will be compared with a single administration of a pain item with a 7-day recall, in order to evaluate if the latter alone is sufficient for measuring pain.
Web-avidity of patients | 6 weeks
  Identify the web-avidity of patients by summarizing patients' responses to questionnaire items about their use of internet and email.

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Basch, MD, Principal Investigator — University of North Carolina
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Washington, Seattle, Washington

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center website — http://unclineberger.org/
- See also: National Cancer Institute (NCI) website — http://www.cancer.gov/